CLINICAL TRIAL: NCT06755112
Title: A Study With Biophysical Methods and Skin Biopsies to Evaluate the Effect on the Skin of Healthy Volunteers of Cosmetic Creams Before and After the Use of Nd:YAG Laser
Brief Title: Efficacy Processes of Aesthetic and Cosmetic Methods
Acronym: EPACM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Vasiliki Gardiki, Laboratory Teaching Stuff, Phd candidate, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 37942/11-05-2021
Record Dates: First submitted 2024-12-22; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Olea europaea stem cells; epilation; skin biopsies; efficacy; biophysical measurements; skin care; formulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo cream (Placebo Comparator): everyday using of placebo cream
  Interventions: Other: Placebo cream
- active cream (Active Comparator): everyday using of active cream
  Interventions: Other: active cream

INTERVENTIONS:
Other: Placebo cream — Placebo cream application
  Arms: placebo cream
Other: active cream — Active cream application
  Arms: active cream

SUMMARY:
Study with biophysical methods and skin biopsies to evaluate the effect on the skin of healthy volunteers of

1. cosmetic creams of Unisooth EG-28® mixture before and after Nd:YAG and
2. the Unisooth EG-28® ingredient with iontophoresis and external application of cosmetic cream with active ingredient Olea vitae PLF®.

OBJECTIVE: To be investigated by approved non-invasive biophysical methods (Directive 2003/15/EC of the European Parliament and of the Council of 27 February 2003 amending Council Directive 76/768/EEC on the approximation of the laws of the Member States relating to cosmetic products. Official Journal L 066, 11/03/2003 P. 0026 - 0035), such as transdermal water loss, erythema, pigmentation, keratin hydration (MPA 5 device), elasticity (Cutometer 575 device) and skin microtopography-thin line skin surface imaging (Skin Visoscan VC 98 and Skin Visiometer) and by minimally invasive methods such as skin biopsies, the effect on the skin of substances with a) anti-inflammatory action and b) antioxidant-anti-ageing action incorporated in cosmetic products when applied alone and/or in combination with other aesthetic approved methods with or without the use of devices used in Aesthetics such as Laser Nd:YAG, or diode laser, iontophoresis.

DETAILED DESCRIPTION:
Background and study aims This study aims to evaluate the effects of certain cosmetic creams on the skin of healthy volunteers. Researchers will use biophysical methods and skin biopsies to assess the impact of these creams, both alone or/and in combination with laser treatments.

The study will include efficacy tests (efficacy tests-claim substantiation) with biophysical methods in healthy volunteers of the above-mentioned bioactive substances incorporated in products when applied on their skin either with topical application or in combination with the use of machinery (iontophoresis) and the comparison of results between the methods used.

Healthy male and female volunteers aged 18 to 65 years can participate in this study. Participants will apply either an active cream or a placebo cream to the inner surface of both arms twice daily (morning and evening) for a certain period. The study will measure transdermal water loss, erythema, pigmentation, and keratin hydration using the MPA 5 device before the beginning of the trial and at the end . Elasticity will be measured using the Cutometer 575 device at the same time points. Additionally, small skin biopsies will be taken before starting the cream application and after 14 days to assess collagen improvement.

The study aims to demonstrate the effectiveness of the active ingredients in the cosmetic formulations. The results will help understand how these ingredients and treatments affect the skin. While the non-invasive tests are safe, the skin biopsies are minimally invasive and carry a small risk of discomfort or minor complications.

Study was conducted at the Established Laboratory of Chemistry - Biochemistry - Cosmetology, Department of Biomedical Sciences, University of West Athens, Aegaleo Alsace Campus (Greece)

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer individuals aged 18 to 65 years, either sex
2. Written and informed consent
3. Healthy volunteers without skin disease or any other diseases (acute or chronic)

Exclusion Criteria:

1. Pregnancy, lactating, or planned pregnancy
2. People who use external application containing steroids for the treatment of skin disease more than one month
3. Participated in the same trial within six months from the interview
4. People with hypersensitive skin
5. Skin abnormalities such as severe acne, erythema, telangiectasia on the test site
6. Used the same or similar cosmetic (or pharmaceutical) on the test site within three months from the interview
7. Have peeling of skin or wrinkles removed within six months from the interview
8. Other unsuitable reasons for clinical trial based on the discretion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss (TEWL) | 2 weeks
  Tewameter MPA-5 Courage + Khazaka electronic GmbH (Germany) was used
keratin hydration | 2 weeks
  Corneometer CM 825 Courage + Khazaka electronic GmbH (Germany) was used
melanin and skin erythema. | 2 weeks
  Mexameter MPA-5 Courage + Khazaka electronic GmbH (Germany) was used
skin elasticity | 2 weeks
  Cutometer MPA 580, Courage + Khazaka electronic GmbH (Germany) was used for skin elasticity parameters: R2: visco-elasticity in % (resistance to the mechanical force versus ability of recovery), R5: net elasticity in %: Ur/Ue = elastic part of the suction phase vs. immediate recovery during relaxation phase, R7: Ur/Uf proportion of the immediate recovery compared to the amplitude after suction in %.
Skin Biopsies | 2 weeks
  Skin puncture biopsies (2.5-3.0 mm) were taken from the forearm of each volunteer. The samples were taken before treatment (Pre-treatment) D=0 and 14 days after laser and product application (Post treatment) D= 14, to all 12 volun-teers. The skin was cleaned with a providone-iodine solution, before taking the biopsy, and the area was anesthetized with a xylocaine solution with epineph-rine. A special cylindrical tool was used, which was rotated through the skin, to remove a small part of the skin, including deeper layers. The incision depth was up to the dermis. The biopsies were placed in numbered vials with formalin so-lution and then fixed for observation under the optical microscope. The goal was to observe the possible increase in the thickness of the epidermis, or the dermis, as well as the morphological observation of the structure of the dermis, in terms of collagen and elastin fibers. The dermis' thickness was measured from the start of the dermoepidermal synapse to the end o

SECONDARY OUTCOMES:
self assesment questionnaire | 2 months
  Finally, forty-five female volunteers aged between 18-65 , phototypes II and III, according to Fitzpatrick classification, were included in the self-questionnaire study after the appropriate signed informed consent. The study was conducted during the years 2022-2023. Treated areas with active cream or placebo were left or right arm, randomly assigned .

CONTACTS AND LOCATIONS:
Overall Officials: ATHANASIA VARVARESOU, PROFESSOR, Study Director — UNIWA
Locations (1):
- UNIWA, Aigáleo, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
University policy